CLINICAL TRIAL: NCT05059002
Title: EpiWatch: Evaluation of a Non-EEG Physiological Signal Based Seizure Monitoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EpiWatch, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EPW001
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-05

CONDITIONS: Epilepsy, Tonic-Clonic
Keywords: Seizure Detection; Seizure; Digital Health
MeSH Terms: conditions — Epilepsy, Tonic-Clonic; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Monitored Subjects (Other): Single arm study of subjects that have been issued an EpIWatch
  Interventions: Device: Physiological signal monitoring and seizure detection

INTERVENTIONS:
Device: Physiological signal monitoring and seizure detection — Data collection and as an adjunct to other methods of seizure monitoring

SUMMARY:
To demonstrate the safety and effectiveness of the EpiWatch device in identifying tonic-clonic (TC) seizures, notifying a third-party of TC seizure occurrence, and collecting non-EEG physiological data for subsequent review during patient hospitalization in an epilepsy monitoring unit (EMU).

DETAILED DESCRIPTION:
To demonstrate the safety and effectiveness of the EpiWatch device in identifying tonic-clonic (TC) seizures, notifying a third-party of TC seizure occurrence, and collecting non-EEG physiological data for subsequent review, during patient hospitalization in an epilepsy monitoring unit (EMU).

Eligible subjects will be issued an EpiWatch device upon admittance into the EMU. The events detected by the EpiWatch will be compared to TC seizures as determined by epileptologists' interpretation of video-EEG recorded for the subject to determine the effectiveness of EpiWatch in detecting TC seizures. EMU standard care practices will not be modified for subjects.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a site EMU for video-EEG monitoring
* Age five and older at the time of enrollment
* Has a clinical history of tonic-clonic (TC) seizures or potential for TC seizures
* Willing and able to comply with study procedures

Exclusion Criteria:

* Has participated previously in EpiWatch development studies or contributed any data to the prior development or evaluation of the detector being tested or previous detectors
* Has any condition that would prevent proper wearing of the watch, its free movement during a seizure, or create discomfort from wearing the watch
* Inability or unwillingness to comply with study procedures

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Comparison of video-EEG to EpiWatch Results for PPA | 6 months
  Lower bound of 95% confidence interval of the positive percent agreement (PPA) > 80%, as determined by comparison to subject video-EEG events as adjudicated based on majority rule of three independent expert reviewers.
Comparison of video-EEG to EpiWatch results for FAR | 6 months
  Upper bound of 95% confidence interval of the false alarm rate (FAR) <.71, as determined by comparison to subject video-EEG events as adjudicated based on majority rule of three independent expert reviewers.

SECONDARY OUTCOMES:
Pediatric Ambulation Positive Percent Agreement | 6 months
  Estimate the PPA in pediatric participants in ambulation in addition to at rest
Pediatric Ambulation False Alarm Rate | 6 months
  Estimate the False Alarm Rate in pediatric participants in ambulation in addition to rest

CONTACTS AND LOCATIONS:
Overall Officials: Gregory L Krauss, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No